CLINICAL TRIAL: NCT03671993
Title: Clinical Effect Observation for Electrical Pudendal Nerve Stimulation in Treating Urethral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShanghaiIAMM
Record Dates: First submitted 2018-09-04; First posted 2018-09-14 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2018-09

CONDITIONS: Pelvic Pain Syndrome
Keywords: urethral pain syndrome; electrical pudendal nerve stimulation; intravesical instillation
MeSH Terms: interventions — Administration, Intravesical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPNS group (Experimental): Electrical pudendal nerve stimulation (EPNS) is a type of conservative treatment which can directly modulate the pudendal nerve and produce a regulation effects on both the sensory fibers and the motor fibers of pudendal nerve.
  Interventions: Procedure: Electrical pudendal nerve stimulation
- II group (Active Comparator): Intravesical instillation (II) are mixture solution administered due to poor oral bio-availability establishing high drug concentrations within the bladder, with few systemic side-effects.
  Interventions: Procedure: Intravesical instillation

INTERVENTIONS:
Procedure: Electrical pudendal nerve stimulation — Four sacrococcygeal points were selected. Two 0.40Х100 mm needles were inserted perpendicularly to a depth of 80-90 mm 1 cm bilateral to the sacrococcygeal joint, to produce a sensation referred to the root of the penis (perineum) or the anus. Two needles of 0.40Х100 or 125mm were inserted obliquely toward the ischiorectal fossa to a depth of 90 to 110 mm about 1 cm bilateral to the tip of the coccyx, to produce a sensation referred to the root of the penis (or the perineum). Each two ipsilaterally needles were connected to one electrode from a G6805-2Multi-Purpose Health Device (Shanghai Medical Instruments High-Techno, Shanghai, China), with a frequency of 2.5 Hz and an intensity (45~55 mA). EPNS was given for 60 min a time, 3 sessions per week for 6 weeks.
  Arms: EPNS group
Procedure: Intravesical instillation — The patient should lie on a couch in a lithotomy position after urination. A catheter was passed through the urethra into the bladder and any residual urine should be drained. A mixture of the Cystistat (sodium hyaluronate, 50ml 40mg, Bioniche Teoranta, Ireland) solution and Lidocaine hydrochloride (40mg :20ml, Fangming Pharmacy company, Shangdong, China) is instilled through the catheter into the bladder. The catheter is then withdrawn leaving the mixture solution inside the bladder, retained for as long as possible, ideally at least 30 minutes. The instillation is once weekly for at 6 weeks.
  Arms: II group

SUMMARY:
In this randomized controlled trial, we intend to determine whether electrical pudendal nerve stimulation is more effective than intravesical instillation in urethral pain syndrome.

DETAILED DESCRIPTION:
According to the 2017 edition of European Association of Urology Guideline, there is no specific treatment for urethral pain syndrome (UPS), and it is recommended this type of patients should be treated in a multi-disciplinary and multi-modal program. Since some mechanisms for the development of UPS suggest it may be a form of bladder pain syndrome (BPS) due to the intimate relation of the urethra with the bladder (both covered with urothelium), a combination of intravesical hyaluronic acid and lidocaine plus sodium bicarbonate, the more widely used regimen for BPS in China, is also applied to UPS here in China. However, the symptom relief of the intravesical irrigation won't last long and patients usually report recurrence in 2-3 weeks. Hence, the purpose of this study is to explore whether the electrical pudendal nerve stimulation（EPNS）, which has been proven effective in treating BPS, is more effective than intravesical instillation (intravesical hyaluronic acid and lidocaine plus sodium bicarbonate) in patients with UPS.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patients aged 18 - 75
2. Occurrence of chronic or recurrent episodic pain perceived in the urethra, especially related to micturition, for more than 3 months; accompanied by other symptoms such as increased daytime and night-time frequency, in the absence of proven infection or other obvious urethral pathology such as urethral diverticulum.
3. Negative in urine routine test or urine cultivation.
4. agreement to sign the written informed consent.

Exclusion Criteria:

1. Symptoms relieved by anti-inflammatory drugs, α-blockers, muscle relaxants.
2. A diagnosis of bacterial cystitis or prostatitis within a 3-month period; bladder or ureteral calculi; active genital herpes; any type of cystitis; vaginitis.
3. life threatening complication such as uterine, cervical, vaginal, or urethral cancer, bladder tumor, heart failure, cardiovascular disease, hemorrhagic disease, uncontrolled diabetes, and/or factors that can affect hemostasis.
4. Female patients with pregnancy or lactation.
5. Serious mental disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Pelvic Pain, Urgency and Frequency Questionnaire ( PUF questionnaire) | 6 weeks
  This instrument consists of eight items that cover areas of pain, urgency, urinary frequency, and symptoms associated with sexual intercourse. The score ranges from 0 to 35 points. Each participant will be evaluated by using the PUF at baseline, three weeks after the treatment commencement and six weeks after the treatment commencement, and we are about to record the mean change of the overall score of this questionnaire.

SECONDARY OUTCOMES:
Visual Analogue Scale for pain | 6 weeks
  Participants will be asked to mark the degree of pain in urethral on a 10-mm VAS, with "0" indicating no pain and "10" indicating the worst painimaginable. Each participant will be evaluated by using this instrument at baseline, three weeks after the treatment commencement and six weeks after the treatment commencement, and we are about to record the mean change of the score.

CONTACTS AND LOCATIONS:
Overall Officials: Siyou Wang, Study Director — Shanghai research institute of acupuncture and meridian
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li T, Feng XY, Feng XM, Lv JW, Lv TT, Wang SY. The short-term efficacy of electrical pudendal nerve stimulation versus intravesical instillation for the urethral pain syndrome: a randomized clinical trial. World J Urol. 2021 Oct;39(10):3993-3998. doi: 10.1007/s00345-021-03698-2. Epub 2021 May 2. PMID 33934208